CLINICAL TRIAL: NCT04157218
Title: Safety and Efficacy of Combining Thread Lifting With Microfocused Ultrasound for Lifting and Tightening the Face
Brief Title: Thread Lifting and Microfocused Ultrasound for Face Tightening Ultrasound for Lifting and Tightening the Face
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0352-19-TLV
Record Dates: First submitted 2019-10-16; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Skin Lifting and Tightening

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of three intervention protocols using Excel 2017 (Microsoft, Redmond, WA, USA):
  1. Treatmnet with HIFU and immediately after, the insertion of lifting threads.
  2. Treatmnet with HIFU and 6 months later, the insertion of lifting threads.
  3. Treatmnet with lifting threads alone .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment with HIFU and immediately after insertion of threads (Active Comparator)
  Interventions: Device: HIFU device (Doublo, HIRONIC Co., Sungnam, Korea); Device: Threads used in this study are absorbable Aptos
- Treatment with HIFU and 6 months later insertion of theads (Active Comparator)
  Interventions: Device: HIFU device (Doublo, HIRONIC Co., Sungnam, Korea); Device: Threads used in this study are absorbable Aptos
- Treatment with lifting threads alone (Active Comparator)
  Interventions: Device: Threads used in this study are absorbable Aptos

INTERVENTIONS:
Device: HIFU device (Doublo, HIRONIC Co., Sungnam, Korea) — The areas treated with HIFU will include: The forehead, temples, and malar area, cheeks and submental area .
  Arms: Treatment with HIFU and 6 months later insertion of theads; Treatment with HIFU and immediately after insertion of threads
Device: Threads used in this study are absorbable Aptos — The threads will be inserted to the cheeks

SUMMARY:
Skin aging is a continuous and inevitable presses usually starting at the age of mid-twenties, this prosses affects all facial layers including skin, subcutaneous fat, superficial muscular aponeurotic system (SMAS), deep facia, the retaining ligaments, muscle activity, and even facial bony structure . The clinical outcome of this process causes the aging signs of the face and neck, including loose facial skin, sagging cheeks, excess skin hanging from the lower jawline and excess fat in the neck .

In the last decade with the introduction of absorbable threads, thread lifting has gained interest and popularity among patients and physicians, as noninvasive technique to treat ptotic skin and reposition of ptotic soft tissue into a more anatomical direction. Histopathological studies indicated that dermal and subcutaneous foreign body reaction after inserting the threads, in forms of collagen deposition, and fibrosis , could explain the tightening effect throughout contracture and remodeling. However, some studies question efficacy especially in the aspects of durability and patient satisfaction .

Another nonsurgical alternative for facial rejuvenation is high-intensity focused ultrasound (HIFU) therapy, during the past decade, HIFU has been used as a clinical noninvasive surgical tool to treat tumors, including those of the liver, prostate, and uterus (10-12) The HIFU devices heat tissue with acoustic energy in a focused, controlled manner. The thermal injury within the tissue leads to focal necrosis and cellular damage, initiating an inflammatory cascade that culminates in tissue remodeling, similar to changes that occur after ablative or nonablative laser treatments .

The Investigators hypothesis that the HIFU treatment followed immediately by thread insertion can amplify and enhance the skin fibrosis, tissue lifting capacity and might give better and longer clinical results in treating ptotic skin.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals.
2. Ages ≥ 30 y.o.
3. Male and female
4. Mild to moderate facial laxity and skin ptosis (Modified Fitzpatrick Wrinkle Scale class 1 and 2 )

Exclusion Criteria:

1. pregnancy
2. breastfeeding,
3. Immunosuppressed individual or individual taking immunosuppressive medications.
4. active systemic or local infections E) collagen vascular disease F) scaring in the planed treatment area G) History of vascular or bleeding disorders H) psychiatric illness I) inability to provide informed consent J) ablative or non-ablative skin procedures in the last 6 months K) surgical procedures within a year to the proposed treatment sites L) Excessive skin laxity on the lower face and neck

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-11-15 (Estimated); Primary Completion 2020-11-15 (Estimated); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in Investigator Global Aesthetic Improvement Scale from baseline to 6 months, and 12 months after treatment for each side of the face | 3, 6 months and 12 months after treatment
  Investigator Global Aesthetic Improvement Scale (IGAIS) from the standardized photographs (0 = no change; 1 = mild improvement; 2 = moderate improve- ment; and 3 = significant improvement)
Change in Subject Global Aesthetic Improvement Scale from baseline to 6 months, and 12 months after treatment for each side of the face. | 3, 6 months and 12 months after treatment
  Subject Global Aesthetic Improvement Scale (SGAIS): (0 = no change; 1 = mild changes; 2 = moderate changes; 3 = significant changes)
Skin lifting in upper, mid and lower part of the face: 3, 6 months and 12 months after treatment for each side of the face | 3, 6 months and 12 months after treatment
  For assessment of skin lifting, the face will be devided into three segmnets : upper, mid, and lower third. The mid-third face-lift will be evaluated by mid-cheek angle. The lower third face-lift will be evaluated by submental lift. The mid-cheek angle will the angle between a horizontal line drawn from alae nasi and a line drawn from alae nasi to the malar prominence.
Wrinkle score, Texture score and pore score calculated by VISIA Software 3, 6 months and 12 months after treatment for each side of the face | 3, 6 months

SECONDARY OUTCOMES:
Occurrence of treatment-related adverse effects collected during the treatment and follow-up periods. | 12 months
  including pain, nerve irritation , numbness/paresthesia , lumps , erythema, tingling, swelling , headache , rash, and pruritus
Patients pain sensation during the treatment for each side of the face at the first visit | 1 month
  Visual Analogue Scale (VAS) (0-10), with 0 denoting no sensation and 10 denoting the worst possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Meical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No